CLINICAL TRIAL: NCT04069195
Title: Placebo Controlled Trial of Docosahexaenoic Acid (DHA) Supplementation in High Risk Pregnancies
Brief Title: Docosahexaenoic Acid (DHA) Supplementation in High Risk Pregnancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH); DSM Nutritional Products, Inc. (Industry); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WRNMMC-2018-0126
Record Dates: First submitted 2018-02-13; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Inflammation; Pregnancy Related
Keywords: Inflammation; DHA; Pregnancy; preterm; overweight
MeSH Terms: conditions — Inflammation; Premature Birth; Overweight | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Double Blinded, Randomized, Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded, randomized, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA supplement (Active Comparator): Patients in the intervention group will recieve a ~1000mg capsule containing ~400mg of DHA. This is not standard of care and is being done for research purposes only. Patients will take this capsule once daily begining between 8-14 weeks of pregnancy until delivery of their infant.
  Interventions: Dietary Supplement: DHA supplement
- corn oil: Soybean oil placebo (Placebo Comparator): Patients in the Placebo group will recieve a ~1000mg capusle containing no DHA and filled with 50:50 mix of corn and soybean oils. This oil is ubiquitous in the american diet and only a very small amount of additional oil will be ingested for study purposes. Giving pregnant women this oil is not standard of care and is being done for research purposes only. Patients will continue taking this placebo from enrollment at 8-14 weeks of pregnancy until time of delivery.
  Interventions: Dietary Supplement: Corn Oil: Soybean Oil

INTERVENTIONS:
Dietary Supplement: DHA supplement — Patient's will be randomized to recieve either DHA or 50:50 corn oil/soybean oil supplement as a once daily supplement to be taken from enrollment through delivery of their infant
  Other Names: Docosahexaenoic Acid
  Arms: DHA supplement
Dietary Supplement: Corn Oil: Soybean Oil — Patient's will be randomized to recieve either DHA or 50:50 corn oil/soybean oil supplement as a once daily supplement to be taken from enrollment through
  Arms: corn oil: Soybean oil placebo

SUMMARY:
Purpose: Determine the effects of maternal docosahexaenoic acid (DHA) supplementation during pregnancy on levels of DHA, synaptamide (novel anti-inflammatory metabolite), and inflammatory biomarkers during pregnancy and at delivery

Research Design: Double blind randomized placebo-controlled study of maternal DHA supplementation during pregnancy.

Methodology /Technical Approach: Investigators plan to enroll 100 pregnant women with a high risk pregnancy related to (1) a pre-pregnancy Body Mass Index (BMI) of ≥30.0 kg/m2 and/or (2) a history of prior preterm delivery at ≤35+6 weeks gestation. Women will be enrolled between the 8th and 14th week of pregnancy and randomized to receive a once daily DHA supplement (DSM Nutritional Products, Columbia Maryland, DHA capsule 441mg/cap) or a placebo (DSM Nutritional Products, Columbia Maryland, Corn Oil/Soybean oil 50/50 mix) for the duration of the pregnancy. DHA is an omega-3 long chain polyunsaturated fatty acid (LCPUFA) and placebo composed of omega-6 LCPUFA's. Investigators will measure maternal levels of plasma DHA, Synaptamide and inflammatory biomarkers at enrollment, at 26-30 weeks of pregnancy, and from cord blood at delivery. Sociodemographic and clinical characteristics will be collected for each mother from pregnancy onset until discharge following delivery. The infant health record and parental report will be reviewed to record clinical data from birth to 12 months corrected age for short term health outcomes potentially related to inflammation-related morbidities, including growth and development, acute infection requiring hospital admission, and any allergic disorder. All plasma samples will be processed at Dr. Kim's NIAAA/NIH laboratories using high-performance liquid chromatography with tandem mass spectrometry

DETAILED DESCRIPTION:
All pregnant women meeting the inclusion/exclusion criteria will be identified at the time of their regular OB appointments between the 8th and the 14th week of pregnancy (+/- 3 days) Research team members will approach potential subjects to explain the study and obtain consent for their participation Patients who give their consent for enrollment will be asked to complete a dietary survey at the time of enrollment Patients will be given a paper script for study drug to be taken to the Walter Reed Military Medical Center pharmacy to obtain study drug The Investigational Pharmacy will randomize the patients in double blinded fashion to the intervention group or placebo group.

Patients in the intervention group will recieve a ~1000mg capsule containing ~400mg of DHA. This is not standard of care and is being done for research purposes only Patients in the Placebo group will recieve a ~1000mg capusle containing no DHA and filled with 50:50 mix of corn and soybean oils. This oil is ubiquitous in the american diet and only a very small amount of additional oil will be ingested for study purposes. Giving pregnant women this oil is not standard of care and is being done for research purposes only The placebo and intervention drugs will be packaged in the same capsule membrane and will be indistinguishable by color, shape, or taste.

Patients will be instructed to take 1 capule PO daily until their child is delivered Patients will be issued a 3 month supply of study drug at enrollment and will get refills from the investigational pharmacy

≤5ml of whole blood will be obtained from each subject at enrollment and at 26-30 weeks gestation (+/- 3 days), as part of a routine blood sampling. It is standard of care to collect blood at this point in pregnancy for lab evaluation. The additional tube of blood collected for this study is for research purposes only and not part of the standard of care. This sample will be centrifuged, and the separated plasma will be labeled and frozen at -80° C pending transport to Dr. Kim's lab at the National Institute on Alcohol Abuse and Alcoholism (NIAAA) for bulk analyses.

At delivery, ≤5ml of umbilical cord blood will be obtained from an umbilical artery and from the umbilical vein. These samples will be processed and stored in a similar fashion as the earlier samples. Cord blood is a medical waste product, and collection will therefore have no adverse effect for either mother or newborn. It is standard of care to collect cord blood by OB request for lab evaluation. Collecting additional cord blood for this study anaylsis is for research purposes only All enrollees will complete a dietary survey upon enrollment at 8-14 weeks (+/- 3 days), at 26-30th week of pregnancy (+/- 3 days), and during the delivery admission. This survey will also include the subject's self-report on compliance with taking the study supplement All plasma samples collected will be processed at Dr. Kim's National Institute on Alcohol Abuse and Alcoholism/ National Insititute of Health (NIAAA/NIH) laboratories The Cytokine Assays for IL-6, Il-10, TNF- alpha will be run in Dr Kim's lab using Ensyme Linked Immunosorbent Assay (ELISA) testing The DHA and Synaptamide levels will be analyzed in Dr. Kim's lab using High performance liquid chromatrography with tandem mass spectrometry All babies from multiple birth pregnancies will be enrolled in this study The offspring of enrolled women will be followed through 12 months corrected age to assess the longer term outcomes of study intervention Information will be collected from the maternal medical record at time of enrollment, infant delivery and postpartum discharge.

Information will be collected from the infant medical record at time of birth discharge, and 12 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* regnant female military health care beneficiaries ≥18 years of age
* Between the 8th and 14th week of pregnancy at enrollment
* BMI of ≥30.0 kg/m2 and/or history of previous preterm delivery at <36 weeks gestation
* Planning to deliver at WRNMMC
* DEERS-eligible
* All infants born to mothers enrolled in this study who do not meet any exclusion criteria

Exclusion Criteria:

* Routine use of DHA supplement (including DHA containing prenatal vitamins) and/or fish consumption greater than twice per week
* Women with a fish allergy
* Known major fetal anomaly believed to be lethal
* Maternal treatment for clotting disorder
* Allergy to corn or soybean oils

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Enrolling only pregnant women and their offspring
Enrollment: 210 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure DHA | Sample obtained between 8-14 weeks of pregnancy
  Measurement of maternal plasma DHA using tandem mass spec
Measure DHA | Sample obtained between 26-30 weeks of pregnancy
  Measurement of maternal plasma DHA using tandem mass spec
Measure DHA | Sample obtained from cord blood at time of infant delivery
  Measurement of fetal plasma DHA using tandem mass spec
Measure synaptamide | Sample obtained between 8-14 weeks of pregnancy
  Measurement of maternal plasma synaptamide using tandem mass spec
Measure synaptamide | Sample obtained between 26-30 weeks of pregnancy
  Measurement of maternal plasma synaptamide using tandem mass spec
Measure synaptamide | Sample obtained from cord blood at time of infant delivery
  Measurement of fetal plasma synaptamide using tandem mass spec
Measure inflammatory biomarkers | Sample obtained between 8-14 weeks of pregnancy
  Measurement of plasma cytokine levels using ELISA human cytokine panel
Measure inflammatory biomarkers | Sample obtained between 26-30 weeks of pregnancy
  Measurement of plasma cytokine levels using ELISA human cytokine panel
Measure inflammatory biomarkers | Sample obtained from cord blood at time of infant delivery
  Measurement of plasma cytokine levels using ELISA human cytokine panel

SECONDARY OUTCOMES:
Maternal Gestational weight gain at end of pregnancy in placebo vs. DHA supplement groups | At time of infant delivery
  Compare maternal gestational weight gain at the end of pregnancy between intervention and placebo groups
Infant delivery method | At time of infant delivery
  Compare delivery method used to delivery infant between intervention and placebo groups
Delivery complications | at time of infant delivery
  Compare any documented delivery complications between intervention and placebo groups
Maternal death | From enrollment in study at 8-14 weeks of pregnancy until 6 months after infant delivery
  Number of maternal deaths in intervention group vs placebo group
Pre-eclampsia | From enrollment in study at 8-14 weeks of pregnancy until 42 weeks of pregnancy or day of infant delivery, whichever happens first
  Presence or absence of pre-eclampsia in intervention vs placebo groups
chorioamionitis | From enrollment in study at 8-14 weeks of pregnancy until 42 weeks of pregnancy or day of infant delivery, whichever happens first
  Presence or absence of chorioamionitis in intervention vs placebo groups
Gestational Diabetes Melitus | From enrollment in study at 8-14 weeks of pregnancy until 42 weeks of pregnancy or day of infant delivery, whichever happens first
  Presence or absence of Gestational Diabetes Mellitus in intervention vs placebo groups
non-gestational Diabetes mellitus | From enrollment in study at 8-14 weeks of pregnancy until 42 weeks of pregnancy or day of infant delivery, whichever happens first
  Presence or absence of non-Gestational Diabetes Mellitus in intervention vs placebo groups
Preterm Premature Rupture of Membranes | From enrollment in study at 8-14 weeks of pregnancy until 42 weeks of pregnancy or day of infant delivery, whichever happens first
  Presence or absence of Preterm Premature Rupture of Membranes in intervention vs placebo groups
going past due dates | during last month of pregnancy
  Presence or absence of going past due dates in intervention vs placebo groups
Placental pathology | at time of delivery
  Any placental pathology documented on maternal delivery summary in intervention vs. placebo groups
Head circumference at birth | At time of infant birth
  Measurement of head circumference at birth in placebo vs. Intervention
Length at birth | At time of infant birth
  Measurement of length at birth in placebo vs. Intervention
weight at birth | At time of infant birth
  Measurement of weight at birth in placebo vs. Intervention
Gestational age at birth | At time of infant birth
  Gestational age at infant birth in both placebo and intervention groups
APGAR score at 1 min | At time of infant birth
  APGAR score assessed for infants in both placebo and intervention groups
APGAR score at 5 min | At time of infant birth
  APGAR score assessed for infants in both placebo and intervention groups
Resuscitation beyond warm/dry stimulate at birth | At time of infant birth
  Presence or absence of any resuscitation beyond warm, dry and stimulate at infant birth
Presence or absence or requirement for respiratory assistance within the first 24 hours after birth | From NICU admission to 24 hours after birth
  Presence or absence of any respiratory support outside of the delivery room in first 24 hours of birth placebo vs intervention groups
Days of antibiotic exposure during birth hospitalization | During birth admission up to 8 months of chronologic age or discharge from hospital whichever happens sooner
  Number of 24hr periods in which infant was exposed to antibiotics during birth hospitalization
NICU admission | Within the first 5 days of infant's life
  Presence or absence of NICU admission in placebo vs intervention groups
Duration of birth admission | Birth through 12 months of age or infant discharge, whichever occurs sooner
  Number of 24hr periods patient was present in hospital during birth admission
Requirement for phototherapy during birth admission | Birth through 14 days of infant life
  Presence or absence of phototherapy during birth admission in placebo vs intervention groups
Culture proven sepsis | From birth through 12 months or until infant discharge whichever occurs sooner
  Presence or absence of culture proven sepsis during birth admission in placebo vs intervention groups
Infant Death | From birth through 12 months or until infant discharge whichever occurs sooner
  Number of infants that died during birth hospitalization in both the placebo and intervention groups
Weight at infant hospital discharge | At time of infant's first discharge from hospital or at 12 months corrected, whichever comes first
  Weight at infant hospital discharge in placebo vs intervention group
head circumference at infant hospital discharge | At time of infant's first discharge from hospital or at 12 months corrected, whichever comes first
  head circumference at infant hospital discharge in placebo vs intervention group
Length at infant hospital discharge | At time of infant's first discharge from hospital or at 12 months corrected, whichever comes first
  Length at infant hospital discharge in placebo vs intervention group
Feeding plan at infant discharge | At 12 months chronological if still admitted or at infant discharge, whichever occurs sooner
  Feeding plan documented as exclusive breastfeeding, formula and breastfeeding or exclusive formula feeding
Infant diagnosis in medical record | at 12 months corrected
  Compare infant diagnosis recorded in medical record in placebo vs intervention group
infant weight at 6 months corrected age | at 6 months corrected
  Weight at 6 months corrected age documented in medical record in placebo vs intervention group
infant weight at 12 months corrected age | at 12 months corrected
  Weight at 12 months corrected age documented in medical record in placebo vs intervention group
head circumferene weight at 6 months corrected age | at 6 months corrected
  head circumferene at 6 months corrected age documented in medical record in placebo vs intervention group
head circumference weight at 12 months corrected age | at 12 months corrected
  head circumference at 12 months corrected age documented in medical record in placebo vs intervention group
Length weight at 6 months corrected age | at 6 months corrected
  Length at 6 months corrected age documented in medical record in placebo vs intervention group
Length weight at 12 months corrected age | at 12 months corrected
  Length at 12 months corrected age documented in medical record in placebo vs intervention group
Number of outpatient visits for infant during first 12 months corrected | birth through12 months corrected
  Number of outpatient visits recorded during first 12 months corrected in placebo vs. intervention groups
Failure to thrive in for infant | birth through 12 months corrected
  Presence or absence of diagnosis "failure to thrive" in medical record through first 12 months corrected in placebo vs intervention
number of inpatient days for infant through 12 months corrected | birth through 12 months corrected
  number of inpatient days for infant through 12 months corrected in intervention vs placebo
Indication of infant developmental delay in medical record from birth through 12 months corrected | birth through 12 months corrected
  Presence or absence of any indication of developmental delay recorded by physician in the medical record through 12 months corrected in intervention vs placebo groups
Number of antibiotic prescriptions for infant through first 12 months corrected | birth through 12 months corrected
  Number of antibiotic prescriptions for infant through first 12 months corrected in intervention vs placebo
Documented infant feeding plan through first year | birth through 12 months corrected
  Documented infant feeding plan through first year. Exclusive breastfeeding, formula and breastfeeding or exclusive formula

CONTACTS AND LOCATIONS:
Overall Officials: Peter F Knickerbocker, DO, Principal Investigator — Walter Reed National Miltary Medical Center; Kim Hee-Yong, PhD, Study Director — NIH/ NIAAA; Carl Hunt, MD, Study Chair — Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed National Miltiary medical center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be coded and master key will only be available to study personnel at Walter Reed National Military Medical Center. No decoded study data will be provided to the NIH/NIAAA

REFERENCES:
- [Background] Valentine CJ. Maternal dietary DHA supplementation to improve inflammatory outcomes in the preterm infant. Adv Nutr. 2012 May 1;3(3):370-6. doi: 10.3945/an.111.001248. PMID 22585914
- [Background] Martin CR, Dasilva DA, Cluette-Brown JE, Dimonda C, Hamill A, Bhutta AQ, Coronel E, Wilschanski M, Stephens AJ, Driscoll DF, Bistrian BR, Ware JH, Zaman MM, Freedman SD. Decreased postnatal docosahexaenoic and arachidonic acid blood levels in premature infants are associated with neonatal morbidities. J Pediatr. 2011 Nov;159(5):743-749.e1-2. doi: 10.1016/j.jpeds.2011.04.039. Epub 2011 Jun 12. PMID 21658712
- [Background] Ma L, Li N, Liu X, Shaw L, Li Calzi S, Grant MB, Neu J. Arginyl-glutamine dipeptide or docosahexaenoic acid attenuate hyperoxia-induced lung injury in neonatal mice. Nutrition. 2012 Nov-Dec;28(11-12):1186-91. doi: 10.1016/j.nut.2012.04.001. PMID 23044165
- [Background] Hofer N, Kothari R, Morris N, Muller W, Resch B. The fetal inflammatory response syndrome is a risk factor for morbidity in preterm neonates. Am J Obstet Gynecol. 2013 Dec;209(6):542.e1-542.e11. doi: 10.1016/j.ajog.2013.08.030. Epub 2013 Aug 29. PMID 23994220
- [Background] De Dooy JJ, Mahieu LM, Van Bever HP. The role of inflammation in the development of chronic lung disease in neonates. Eur J Pediatr. 2001 Aug;160(8):457-63. doi: 10.1007/s004310100785. PMID 11548181
- [Background] Cheng SB, Sharma S. Interleukin-10: a pleiotropic regulator in pregnancy. Am J Reprod Immunol. 2015 Jun;73(6):487-500. doi: 10.1111/aji.12329. Epub 2014 Oct 1. PMID 25269386
- [Background] Kim HY, Spector AA. Synaptamide, endocannabinoid-like derivative of docosahexaenoic acid with cannabinoid-independent function. Prostaglandins Leukot Essent Fatty Acids. 2013 Jan;88(1):121-5. doi: 10.1016/j.plefa.2012.08.002. Epub 2012 Sep 5. PMID 22959887
- [Background] Meijerink J, Poland M, Balvers MG, Plastina P, Lute C, Dwarkasing J, van Norren K, Witkamp RF. Inhibition of COX-2-mediated eicosanoid production plays a major role in the anti-inflammatory effects of the endocannabinoid N-docosahexaenoylethanolamine (DHEA) in macrophages. Br J Pharmacol. 2015 Jan;172(1):24-37. doi: 10.1111/bph.12747. Epub 2014 Sep 23. PMID 24780080
- [Background] Balvers MG, Verhoeckx KC, Plastina P, Wortelboer HM, Meijerink J, Witkamp RF. Docosahexaenoic acid and eicosapentaenoic acid are converted by 3T3-L1 adipocytes to N-acyl ethanolamines with anti-inflammatory properties. Biochim Biophys Acta. 2010 Oct;1801(10):1107-14. doi: 10.1016/j.bbalip.2010.06.006. Epub 2010 Jun 27. PMID 20601112
- [Background] Makrides M, Gibson RA, McPhee AJ, Yelland L, Quinlivan J, Ryan P; DOMInO Investigative Team. Effect of DHA supplementation during pregnancy on maternal depression and neurodevelopment of young children: a randomized controlled trial. JAMA. 2010 Oct 20;304(15):1675-83. doi: 10.1001/jama.2010.1507. PMID 20959577
- [Background] Dunstan JA, Simmer K, Dixon G, Prescott SL. Cognitive assessment of children at age 2(1/2) years after maternal fish oil supplementation in pregnancy: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2008 Jan;93(1):F45-50. doi: 10.1136/adc.2006.099085. Epub 2006 Dec 21. PMID 17185423